CLINICAL TRIAL: NCT01577927
Title: Feasibility and Efficacy of a Home Rehabilitative Network for Prolonged Weaned Patients Discharged From a Weaning Unit
Brief Title: Feasibility Study of a Home Rehabilitative Network to Treat Prolonged Weaned Patients
Acronym: UTIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Salvatore Maugeri (Other)
Responsible Party: Principal Investigator, Michele Vitacca, Principal investigator, Fondazione Salvatore Maugeri
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UTIR; Dlg. 5685 on 28 May 2010 (Other Grant/Funding Number: Lombardy Region)
Record Dates: First submitted 2012-04-10; First posted 2012-04-16 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Diseases
Keywords: weaning; severe chronic diseases; UTIR
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual home care (Active Comparator): No assistance or care by PT.
  Interventions: Other: Usual home care
- PT-assisted home rehabilitation (Experimental): Assisted home care is supported by a PT at least 2 times/month. Few brief educational lessons preceeded the training activity that the patient performs by himself at home.
  Interventions: Behavioral: PT-assisted home rehabilitation

INTERVENTIONS:
Other: Usual home care — Usual home care consists in supporting drug and oxygen therapy, mechanical ventilation, GP's assistance,and periodical in-hospital visit.
  Arms: Usual home care
Behavioral: PT-assisted home rehabilitation — Patient performs 50 min physical activity/working day autonomously by the help of a DVD. The physical activity consists in cyclette, calisthenic exercises, and training of the respiratory muscles.
  Every two weeks, PT phones the patient for an educational reinforcement.
  Arms: PT-assisted home rehabilitation

SUMMARY:
Patients at high complexity with severe chronic diseases can require several admission in intensive care units (ICU) to overcome acute exacerbations by the use of assisted ventilation. In the last 10 years, new technologies and beds in ICU evidenced a new group of patients often needing weaning procedures due to a long-lasting period of mechanical ventilation. These patients are often under chronic conditions with recurrent symptoms, reduced effort tolerance and depression.

Weaning process is a frail step in the medical history of a patient who has survived an acute episode of respiratory failure and has spent a period of time under mechanical ventilation. Patients are followed for the duration of in-hospital stay, an expected average period of 4 weeks.

When discharged fron an Intensive Care Unit (ICU) or a weaning center, the patient is usually managed by GPs and by the hospital where he has been admitted to following re-exacerbations. The conventional approach is for sure inadequate for this type of patient whose clinical complexity, disability and frailty need for a continuity of care through a higher complex approach of management.

A structured program of Home Rehabilitation could be a possible solution to this problem. Thus, the hypothesis of the study is to evaluate feasibility and sustainability and efficacy of a home rehabilitative network for prolonged weaned patients discharged from a weaning unit.

DETAILED DESCRIPTION:
Patients referred to the Fondazione Salvatore Maugeri for prolonged weaning are enrolled and trained in an individualised program of home care in order to recover their own autonomies. Home care compares 2 arms: usual care vs physiotherapist (PT)-assisted care. Usual care consists in supporting drug and oxygen therapy, mechanical ventilation, GP's assistance, periodical in-hospital visit. The PT-assisted home care is supported by PT at least 2 times/month, autonomous 50 min physical activity/working day by the help of a DVD. The physical activity consists in cyclette, calisthenic exercises, and training of the respiratory muscles. Few brief educational lessons by PT preceded the training activity. Every two weeks, PT calls the patient by phone for an educational reinforcement.

ELIGIBILITY:
* General Inclusion criteria: 1. Signature of the informed 2. Good expectation of life
* Specific Inclusion Criteria : Score of general dependences < 19 according to the Critical Patients Autonomy Planning (CPAP) Scale

Exclusion Criteria:

* Patient with neuromuscular, highly progressive neurological diseases (i.e. amyotrophic lateral sclerosis), patient requiring surgical interventions, sedation, and hemodialysis.
* Unstable patient conditions as daily variability of the blood arterial pressure >20%, arrhythmias, PaO2/FiO2 < 300, unsatisfactory respiratory pattern, haemoglobin < 7 g /dL, temperature > 38°C, presence of neurological or orthopaedic side effects, and recent embolisms from TVP. Refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-07; Primary Completion 2013-01 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Critical Patients Autonomy Planning (CPAP) | Changes from baseline and 4 weeks, and 6 months after home activity
  CPAP is a measure of dependency. CPAP was evaluated at three different time-points: at in-hospital admission (baseline), at discharge (patients are followed for the duration of their in-hospital stay, an expected average time of 4 weeks), and after 6 months of physical activity at home.

SECONDARY OUTCOMES:
Maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP) | Changes from baseline and 4 weeks (average time), and 6 months after home activity
  Respiratory Functionality
MRF 26 | Changes between discharge at 4 weeks (average time) and 6 months after home activity
  Quality of life evaluation.
Likert Scale | Changes between discharge at 4 weeks (average time) and 6 months after home activity
  Satisfaction for patient/caregiver
Mortality | Changes between 3, 6 and 12 months post-discharge
  Clinical measure
MRC Scale and/or dynamometer | Changes between baseline, discharge at 4 weeks, and 6 months after home activity
  Rehabilitative measure referring to muscles force
6-min walking test | Changes from baseline and discharge at 4 weeks, and 6 months after home activity
  Rehabilitative measure evaluating the effort tolerance.
EuroQol | Changes between discharge at 4 weeks (average time) and 6 months after home activity
  Quality of life evaluation
Gussago Nursing Scale | Changes from baseline and 4 weeks, and 6 months after home activity
  Measure of dependency.
Barthel Index | Changes from baseline and 4 weeks, and 6 months after home activity
  Measure of dependency.
Pre-morbidity life-style (PLS) | Changes from baseline and 4 weeks, and 6 months after home activity
  Measure of dependency.

CONTACTS AND LOCATIONS:
Overall Officials: Piero Ceriana, MD, Principal Investigator — Fondazione Salvatore Maugeri; Michele Vitacca, MD, Study Director — Fondazione Salvatore Maugeri
Locations (1):
- Fondazione Salvatore Maugeri, Lumezzane, Brescia, Italy

REFERENCES:
- [Derived] Vitacca M, Barbano L, Vanoglio F, Luisa A, Bernocchi P, Giordano A, Paneroni M. Does 6-Month Home Caregiver-Supervised Physiotherapy Improve Post-Critical Care Outcomes?: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2016 Aug;95(8):571-9. doi: 10.1097/PHM.0000000000000441. PMID 26829083